CLINICAL TRIAL: NCT02845414
Title: Phase I Study Of Stem-Cell Directed Deimmunized CD133KDEL Toxin In The Treatment Of Solid Tumors
Brief Title: Study of CD133KDEL Toxin in the Treatment for Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016LS026
Record Dates: First submitted 2016-07-18; First posted 2016-07-27 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intravenous Infusion of dCD133KDEL (Experimental)
  Interventions: Drug: CD133KDEL (dCD133KDEL)

INTERVENTIONS:
Drug: CD133KDEL (dCD133KDEL) — Patients will receive dCD133KDEL at the assigned dose level via a 30-minute intravenous infusion on days 1, 3, 5, 8, 10 and 12 (total of 6 doses) of a 28-day cycle.

SUMMARY:
This is a single center, phase I dose escalation study designed to determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of deimmunized CD133KDEL (dCD133KDEL), a ligand-directed, deimmunized pseudomonas toxin against CD133, in patients with advanced, previously treated, refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or cytologically confirmed, metastatic or unresectable solid tumor malignancy.
2. Measurable or evaluable disease per RECIST 1.1 criteria (Appendix II), or modified RECIST criteria for mesothelioma (Appendix II).
3. At least 1 prior line of systemic therapy considered standard for the malignancy, and for which no standard therapies exist. Prior systemic chemotherapy, immunotherapy, biological therapy, radiation therapy and/or surgery are allowed before the first dose of dCD133KDEL with the following restrictions:

   * At least 14 days since any systemic therapy.
   * At least 28 days since any experimental therapy.
   * At least 14 days since any radiation therapy.
   * At least 28 days since any major surgery, defined as a surgery involving a risk to the life of the patient, specifically, an operation upon an organ within the cranium, chest, abdomen, or pelvic cavity.
4. Recovered from the acute toxic effects (≤ grade 1, CTCAE v4.0) of previous cancer treatment prior to study registration.
5. ECOG performance status 0 or 1 (Appendix III).
6. Adequate organ function within 14 days of study registration, defined as follows System Parameter Laboratory Value Hematologic Absolute neutrophil count (ANC) ≥1.5 x 10^9 /L Hemoglobin* 9 g/dL Platelets* ≥100 x 10^9 /L Hepatic Total bilirubin < 2 x ULN^ ALT < 2 x ULN^ Renal Serum creatinine < 1.5 mg/dL OR estimated GFR >50 by modified Cockcroft-Gault (* Patient may not have had a transfusion within 7 days

   ^ Upper limit of institutional normal.)
7. Albumin ≥ 3.0 gm/dL within 14 days of study registration.
8. Adequate cardiac function, defined as an ejection fraction ≥40% on transthoracic echocardiogram done within 14 days of study registration.
9. QT/QTc interval ≤ 450 milliseconds within 14 days of study registration. If this screening EKG demonstrates a QT/QTc interval > 450 milliseconds, a second screening EKG will be done within 7 days to document that the QT prolongation is persistent. The patient will be eligible if the second screening EKG shows a QT/QTc interval ≤ 450 milliseconds but will require additional EKGs during the study period as outlined in section 6.1.2.
10. Adequate pulmonary function, defined as resting oxygen saturation ≥ 90% on room air and/or pulmonary function tests (PFT) showing corrected DLCO >50% and FEV1 ≥ 2 liters or ≥ 60% of predicted. PFT testing is required within 28 days of study registration only if the patient is symptomatic or prior known impairment is present.
11. Females of childbearing potential and males who have partners of childbearing potential must agree to use 2 effective contraception methods, one of which must be a barrier method, during the study and for ≥12 weeks after the last dose of dCD133KDEL. Effective methods include intrauterine device (IUD), Depo-Provera injection or implant, Evra patch, NuvaRing, oral contraception, and diaphragm/spermicide with condom.
12. Ability to understand and provide voluntary written consent.

Exclusion Criteria:

1. Known active CNS metastases or neurological symptoms possibly related to CNS metastases, spinal cord compression, or evidence of leptomeningeal disease. Patients with a history of brain metastases who have undergone whole brain radiation or gamma knife treatment ≥ 28 days prior to registration, whose metastases are documented as stable or resolved at the time of screening by brain MRI (or head CT with contrast for those who are intolerant of MRI), and do not require ≥10 mg of prednisone equivalent for symptom management related to the brain metastases, are eligible.
2. Known uncontrolled cardiac arrhythmias, electrocardiographic evidence of acute ischemia or active conduction system abnormalities within 28 days of registration.
3. Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements.
4. History of any one or more cardiovascular conditions within 12 weeks of study registration

   * cardiac angioplasty or stenting
   * myocardial infarction
   * unstable angina
   * coronary artery bypass graft surgery
   * symptomatic peripheral vascular disease
   * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA, Appendix IV)
   * transient ischemic attack and/or cerebrovascular accident
5. History of another malignancy other than non-melanoma skin cancer or treated carcinoma in situ, unless documented to be disease free for at least 3 years.
6. History of allergic reaction or sensitivity to compounds of similar chemical or biological composition to dCD133KDEL, or any of the components of dCD133KDEL (i.e. Polysorbate 80).
7. Pregnant or breastfeeding women, or women intending to become pregnant. Females of child bearing potential must have a negative serum pregnancy test within 14 days of study registration.
8. Prior toxin-directed therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Day 28
  Maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
Dose Limiting Toxicity (DLT) | 21 days after the first dose of dCD133KDEL
  A ≥ grade 3 (CTCAE v4.0) adverse event within 21 days after the first dose of dCD133KDEL and at least possibility attributable to dCD133KDEL
Tumor response defined as partial and complete response according to RECIST 1.1 criteria, with its 95% confidence interval | Disease assessment between days 29, 30, 31, 32, 33. Follow up for disease response every weeks 6, 7 ,8 ,9, 10,11,12
  Tumor response will be evaluated and summarized by dose level in a contingency table with its 95% confidence interval

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Fujioka, MD, Principal Investigator — University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States